CLINICAL TRIAL: NCT04114487
Title: Effect of Dual Task Balance Training on Cognitive Functions in People With Mental Retarded
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ebrar atak, MSc(PT), Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ebraratak
Record Dates: First submitted 2019-08-06; First posted 2019-10-03 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Rehabilitation
Keywords: Cognitive rehabilitation; Dual task; Balance; Motor skills

STUDY DESIGN:
Intervention Model Description: The 45-person study group will be randomized to 3 groups of 15 persons each. The first group will not be subjected to any application except education. The second group will be the control group and will be taken to the balance training in addition to normal education. In the third group, dual task balance training will be applied within the scope of cognitive rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control 1 (No Intervention): The control 1 group will not be subjected to any application except education.
- control 2 (Active Comparator): The control 2 group will be the control group and will be taken to the balance training in addition to normal education.
  Interventions: Other: dual task balance training
- intervention (Experimental): In theintervention group, dual task balance training will be applied within the scope of cognitive rehabilitation.
  Interventions: Other: dual task balance training

INTERVENTIONS:
Other: dual task balance training — The studies were planned to be 2 times a week for 12 weeks. The 20-minute Dual Task balance training program is planned to be composed of two sections of 10 minutes. In the first 10 min section, the individual will exercise with the multi-task mode of CogniBoard on the balance ball. . Stroop study will be performed on the balance ball in the second 10 minutes of the exercise.
  Other Names: classic balance training
  Arms: control 2; intervention

SUMMARY:
With this study, it will be tried to determine whether the addition of physiotherapy program to the education of mentally disabled individuals is effective and necessary in terms of mental performance.

DETAILED DESCRIPTION:
Mental disability levels IQ = 50-79 individuals with mild / border mental disabilities will be included in the study. The disability status of the individuals will be determined by the health report, and the cognitive status of the individuals will be determined by the report given as a result of the evaluation made by the Guidance Research Centers of the National Education Directorates. The 45-person study group will be randomized to 3 groups of 15 persons each. The first group will not be subjected to any application except education. The second group will be the control group and will be taken to the balance training in addition to normal education. In the third group, dual task balance training will be applied within the scope of cognitive rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* IQ 50-79
* 6-14 years old
* take command of Turkish
* do not have physical disability
* not have metabolic and systemic disease
* To have a report on the mental disability and education required by the Ministry of National Education

Exclusion Criteria:

* To have any situation that prevents the taking of commands related to the exercise program to be implemented
* To have a chronic systemic disease
* To have an educational diagnosis other than the mental disability

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
cognitive functions | 3 months
  short-term memory(visual memory test, memorize the squares,number of correct choices), İnformation processing speed (space bar presses in response to non-target stimulus to be impulsive behavior. number of errors), Focusing and Perception (space bar presses in response to a target stimulus.The difference between the number of target stimuli that appeared in the test and the number of correct responses gives the number of omission errors. )

SECONDARY OUTCOMES:
motor functions | 3 months
  balance (walking forward a line, number of steps), coordination(jumping in place-same sides synchronized-number of correct form) , manual dexterity(transferring pennies-number of 15 sec.), gross motor skills and upper-limb coordination (dribling a ball-alternating hands-number of dribbles)

CONTACTS AND LOCATIONS:
Overall Officials: Ebrar Atak, MSc, Principal Investigator — Gerçek Dünya special education and rehabilitation center
Locations (1):
- Ebrar Atak, Yalova, Turkey (Türkiye)

DOCUMENTS (2):
  • Study Protocol (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04114487/Prot_001.pdf
  • Informed Consent Form (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04114487/ICF_000.pdf